CLINICAL TRIAL: NCT03249220
Title: Clinical Pilot Study to Evaluate a New Multi-parameter Neuromonitoring Device That Allows the Measurement of Regional Cerebral Blood Flow (rCBF), Intracranial Pressure (ICP), Brain Temperature Monitoring and Ventricular Cerebrospinal Fluid (CSF) Drainage in Brain-injured Patients
Brief Title: Clinical Pilot Study to Evaluate a New Multi-parameter Neuromonitoring Device in Brain-injured Patients
Acronym: CBMS FIH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carag AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2015.5703
Record Dates: First submitted 2017-08-02; First posted 2017-08-15 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBMS (Experimental)
  Interventions: Device: Placement of the CBMS Probe

INTERVENTIONS:
Device: Placement of the CBMS Probe — Patients will be treated according to standard care in place at the investigation site, when intra-ventricular drainage is needed. Patients will receive the new multifunctional device (CBMS Probe) instead of the single function device generally used. Drainage will be performed by routine standards. Temperature, intracranial pressure and cerebral blood flow will be recorded. Treatment decision will be made by the neurointensive care specialist based on standard care.

SUMMARY:
Clinical pilot study to evaluate a new multi-parameter neuromonitoring device that allows the measurement of regional cerebral blood flow (rCBF), intracranial pressure (ICP), brain temperature monitoring and ventricular cerebrospinal fluid (CSF) drainage in brain-injured patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patient, aged 18 - 75 years
* Brain injured patients with acute intracranial hemorrhage (including aneurysmal subarachnoid hemorrhage (SAH) and spontaneous intracerebral hemorrhage (ICH)) who are admitted to the ICU and have an indication for ICP monitoring and CSF drainage, as per standard patient care
* Informed consent obtained for research in emergency situations according to HRA art. 30 & 31 at time of inclusion

Exclusion Criteria:

* Known kidney disease, defined as plasma creatinine > 120 μmol/l
* Known liver disease, defined as AST > 200 IU/L
* Over-active thyroid or benign tumors of the thyroid
* History of allergic disorders, including allergic reactions, against contrast agents containing iodine, or against ICG
* Patients which have received one of the following medications before being admitted to ICU: Haloperidol, Meperidine, Methadone, Morphine, Phenobarbital and Rifamycin.
* Patients with wounds or scars including the front orbital region.
* Cerebrospinal fluid infection or signs of meningo-encephalitis
* Anemia (hemoglobin < 10 g/dl) or Thalassemia
* Carbon monoxide poisoning
* Acquired pathological or congenital disorders of the cerebral system, being clinically significant, respectively interfering in the investigator's opinion with the conduct of study
* Documented history of bleeding, clotting or coagulation disorders
* Patients who are not suitable for a CT perfusion
* Subjects who, in the opinion of the investigator, will be inappropriate for inclusion into this clinical investigation or will not comply with requirements of the study
* Any disorder in the investigator's opinion that could interfere with compliance of safety evaluation
* Pre-existing disability and/or legal representative
* Patients who are kept lawfully in an institution
* Participation in another interventional clinical investigation within the last 30 days before start of treatment
* History of, respectively diagnosis of pregnancy, or breastfeeding patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Comparability of regional CBF values and values obtained with CT perfusion and TCD | Up to 28 days until probe removal
  Regional CBF values calculated with the investigational devices (CBMS) are within ranges described in literature, and dynamic changes of regional CBF are consistent to those values obtained with established methods CT perfusion and TCD.

SECONDARY OUTCOMES:
Safety related to catheter insertion and monitoring | Until 7 days after probe removal
  Safety related to catheter insertion and monitoring: local hematomas, infections, CSF drainage dysfunction in comparison with other standard intra-ventricular devices.

CONTACTS AND LOCATIONS:
Overall Officials: Werner Z'Graggen, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (2):
- Switzerland (2):
  - Inselspital Bern, Bern, Canton of Bern
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne, Canton of Vaud

IPD SHARING:
Plan to Share IPD: Undecided